CLINICAL TRIAL: NCT02793986
Title: Dexmedetomidine vs Propofol Sedation Reduces Postoperative Delirium in Patients Receiving Hip Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PJ2015-07-12
Record Dates: First submitted 2016-06-04; First posted 2016-06-08 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2016-06

CONDITIONS: Anesthesia; Local Anesthesia
MeSH Terms: interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexmedetomidine sedation (Experimental): Patients received local anesthesia, in this arm, the sedation of patients was achieved with a bolus of dexmedetomidine at 1.0 μg/kg (over a period of 15 to 20 min) and followed by an infusion of dexmedetomidine at 0.2-0.7 μg/kg/h.
  Interventions: Drug: dexmedetomidine
- propofol sedation (Experimental): Patients received local anesthesia, in this arm, the sedation of patients was achieved with a target-controlled infusion (TCI) of propofol, and the effect site concentration was set to 0.8-1.0μg/ml.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — For patients in Group P, the sedation was achieved with a target-controlled infusion (TCI) of propofol, and the effect site concentration was set to 0.8-1.0μg/ml.
  Arms: propofol sedation
Drug: dexmedetomidine — For patients in Group D, the sedation was achieved with a bolus of dexmedetomidine at 1.0 μg/kg (over a period of 15 to 20 min) and followed by an infusion of dexmedetomidine at 0.2-0.7 μg/kg/h. The depth of sedation was considered enough when patient was unresponsive to voice.
  Arms: dexmedetomidine sedation

SUMMARY:
With blocks of lumbar and lumbar plexus, we can reduce the intravenous anesthetics usage. To offer an satisfied surgery process for patients, a proper sedation is necessary. So in this study, we want to investigate the influence of two different sedative drugs on outcomes of patients received hip replacement surgery .

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older and undergoing hip fracture repair

Exclusion Criteria:

* Patients with severe cognitive impairment (MMSE score, <15)
* Preoperative delirium as determined by Confusion Assessment Method
* Contraindications to local anesthesia
* Prior hip surgery
* Mental or language barriers that would preclude data collection
* Severe congestive heart failure (NewYork Heart Association class IV)
* Severe chronic obstructive pulmonary disease (Global Initiative for Chronic Obstructive Lung Disease guidelines, stage III-IV)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 296 (Actual)
Dates: Start 2015-08; Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 7 days after surgery
Mortality in 30 days after surgery | 30 days after surgery

SECONDARY OUTCOMES:
Complications of cardiopulmonary system | 30 days after surgery
Incidence of cerebrovascular accident | 30 days after surgery
Out of bed time | 7 days after surgery
Discharge time | 30 days after surgery
Dosage of vasoactive agent | During sugary
Extubation time | 7 days after surgery
Hemodynamic index | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Gu, PHD, Study Director — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- The first affiliated hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu X, Xie G, Zhang K, Song S, Song F, Jin Y, Fang X. Dexmedetomidine vs propofol sedation reduces delirium in patients after cardiac surgery: A meta-analysis with trial sequential analysis of randomized controlled trials. J Crit Care. 2017 Apr;38:190-196. doi: 10.1016/j.jcrc.2016.10.026. Epub 2016 Nov 11. PMID 27936404
- [Background] Li X, Yang J, Nie XL, Zhang Y, Li XY, Li LH, Wang DX, Ma D. Impact of dexmedetomidine on the incidence of delirium in elderly patients after cardiac surgery: A randomized controlled trial. PLoS One. 2017 Feb 9;12(2):e0170757. doi: 10.1371/journal.pone.0170757. eCollection 2017. PMID 28182690
- [Background] Orena EF, King AB, Hughes CG. The role of anesthesia in the prevention of postoperative delirium: a systematic review. Minerva Anestesiol. 2016 Jun;82(6):669-83. Epub 2016 Jan 28. PMID 26822815
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303